CLINICAL TRIAL: NCT02627937
Title: Clinical Predictors of Pediatric Obstructive Sleep Apnea/Hypopnea Syndrome
Brief Title: Clinical Predictors of Pediatric OSAHS
Acronym: PEDOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGMH IRB NO. 104-3716B
Record Dates: First submitted 2015-11-06; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-10

CONDITIONS: Pediatric Sleep Apnea
Keywords: Pediatric obstructive sleep apnea/hypopnea syndrome; Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pediatric sleep apnea: The children were confirmed to have OSAHS by comprehensive polysomnography (PSG).

SUMMARY:
The purpose of this study is to develop adequate and satisfactory tools using reliable clinical and physical factors in predicting pediatric obstructive sleep apnea/hypopnea syndrome (OSAHS) and allow greater access to appropriate therapy in children.

DETAILED DESCRIPTION:
The prevalence of OSAHS is estimated to be about 1% to 4% in children, however, it is frequently underdiagnosed because of the difficulties for evaluation.Current diagnostic approaches are based on the patient's history, clinical presentation and physical examination, endoscopy, and radiological imaging examinations, and confirmation is made by the current gold standard of full-night polysomnography (PSG). Previous studies have reported the use of a clinical history, physical examination and questionnaires for predicting pediatric OSAHS but there were lacking of adequate and satisfactory results. Despite the potential diagnostic benefits, PSG for pediatric patients are not routinely used in clinical practice. Therefore, to obtain a reliable, valid, and easily-performed diagnostic or screening tool for the clinical assessment of pediatric OSAHS is essential for the cost-effective care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* children (younger than 18 years old and older than 2 years old) with symptoms of snoring and then were confirmed to having obstructive sleep apnea/hypopnea syndrome by a comprehensive polysomnography

Exclusion Criteria:

* patients with substance abuse problems or the long-term usage of medications known to affect sleep, craniofacial abnormalities or neuromuscular disorders, Down syndrome, cerebral palsy, mucopolysaccharidoses, Prader-Willi syndrome, history of psychosis, central sleep apnea syndrome, or previous airway surgery including tonsillectomy and/or adenoidectomy were excluded from the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children with chief complaints of snoring
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Clinical predictors for apnea/hypopnea index (AHI) | up to 4 months
  When all variables were analyzed individually with the AHI, Spearman rank correlation analysis was used to explore the relationships between clinical predictor variables and AHI.Significant variables were entered into stepwise multiple linear regression analysis to identify independent predictors for pediatric OSAHS and to develop a predictive equation for AHI values.

SECONDARY OUTCOMES:
Anthropometric measurements: body mass index z-score (BMI z-score) | up to 4 months
  BMI z-score: a measure of relative weight adjusted for the child's age and gender, and calculated by dividing the difference between the measured value and the mean by the standard deviation.
Anthropometric measurements: tonsil size grading | up to 4 months
  Tonsil size grading: 0, surgically removed tonsils; 1, tonsils hidden within the pillars; 2, tonsils extending to the pillars; 3, tonsils were beyond the pillars but not to the midline; and 4, tonsils extended to the midline.
Anthropometric measurements: modified Mallampati grade (aka updated Friedman's tongue position | up to 4 months
  updated Friedman's tongue position: I: visualization of the entire uvula and tonsils/pillars.; IIa: visualization of most of the uvula, but the tonsils/pillars are absent.; IIb: visualization of the entire soft plate to the base of the uvula.; III: visualization of some of the soft palate, but the distal structures are absent.; IV: visualization of the hard palate only.
Anthropometric measurements: uvular length | up to 4 months
  uvular length in centimeter
Snoring visual analogue scale (Snoring VAS) | up to 4 months
  Snoring VAS (Units on a Scale): 0-10, 0 = "no snoring noise" and 10 = "the loudest sound imaginable
Apnea/hypopnea index (AHI) | up to 4 months
  AHI: total number of apneas and hypopneas per hour of electroencephalographic sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Ching Lin, MD, Principal Investigator — Department of Otolaryngology, Sleep Center, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Department of Otolaryngology, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan, Taiwan